CLINICAL TRIAL: NCT04760184
Title: Impact of COVID-19 on Patients Treated With Autologous Hematopoietic Stem Cell Transplantation in Sweden - a Retrospective Cohort Study
Brief Title: Impact of COVID-19 After Autologous Hematopoietic Stem Cell Transplantation in Sweden
Acronym: AutoCOVID-19
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other); Lund University Hospital (Other); University Hospital, Linkoeping (Other); University Hospital, Umeå (Other); Region Örebro County (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-03433
Record Dates: First submitted 2020-12-11; First posted 2021-02-18 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Myeloma Multiple; Malignant Lymphoma; Hematologic Neoplasms; Stem Cell Transplant Complications
Keywords: Autologous stem cell transplantation; COVID-19
MeSH Terms: conditions — COVID-19; Multiple Myeloma; Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID19 positives after autologous stem cell transplantation: All Swedish citizens treated with ASCT for malignant disease in Sweden from 1st January 2020 until 31st December 2020 who has tested positive for SARS-CoV-2 from start of conditioning until the end of the study period 31st March 2021.
  Interventions: Other: Autologous stem cell transplantation

INTERVENTIONS:
Other: Autologous stem cell transplantation — The study will describe the implications of COVID-19 infection following autologous stem cell transplantation

SUMMARY:
This retrospective observational cohort study aims to describe the impact of COVID-19 in patients treated with autologous stem cell transplantation (ASCT) for malignant disease in terms of risk factors, morbidity, need for supportive care and mortality. All patients treated with ASCT in Sweden from 1st January 2020 until 31st December 2020 are eligible for this study. Patients who also has tested positive for SARS-CoV-2 from start of conditioning or later will be identified through the national registry of the Public Health Agency of Sweden and a systematic analysis of their medical records will be performed.

DETAILED DESCRIPTION:
Research question How does infection with SARS-CoV-2 affect patients with hematological malignancies who are treated with autologous hematopoietic stem cell transplantation?

Study population All Swedish citizens treated with ASCT for malignant disease in Sweden from 1st January 2020 until 31st December 2020 are eligible for this study. There will be a minimum follow-up time of one month for all patients.

Data collection and storage Patients will be identified using local ASCT registers at the seven university hospitals, as there is no national register for ASCT-patients in Sweden. These seven university hospitals are the only sights to perform ASCT in Sweden. The Public Health Agency of Sweden (Folkhälsomyndigheten - FHM) has the national responsibility to surveil and control communicable disease. The FHM uses several different surveillance systems to monitor the spread of COVID-19. Since COVID-19 is subject to mandatory reporting under the Communicable Diseases Act, physicians and laboratories continuously supply data to be analyzed daily by the FHM. The coverage of this database is estimated to be very high, close to 100%. For this study the investigators will link the patients identified through the ASCT-centers with the register of SARS-Cov-2 positive patients (SmiNet) held by the FHM. Patients who has tested positive for SARS-CoV-2 on the day of start of conditioning or at any given time thereafter will be included in the study. Inclusion of positive SARS-CoV-2 tests will start from 1st January 2020 until 31st March 2021 to allow for 3 months of follow-up after transplantation. For every ASCT-patient that has tested positive for COVID-19 after ASCT a systematic analysis of their medical records will be performed to describe the circumstances, impact and outcome of the COVID-19.

All data collected will be stored in a deidentified data set on a secure server held by Dalarna Country Council where name and social security number have been erased and given a coded study number. Each patient will only be identified using a separately stored code key. All storage, correspondence and analysis with the code key and pseudonymized data set will adhere to current European General Data Protection Regulation (GDPR) guidelines. The code key will be destroyed as soon as data collection is completed, data quality is secured and the final report is published. The data set will be stored for 10 years and then be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hematological cancer (C81-C96 according to the International Classification of Diseases 10th revision (ICD-10).
* Autologous hematopoietic stem cell transplantation performed 1 January 2020 until 31st December 2020 at a Swedish transplantation center.
* Positive RT-PCR test for SARS-CoV-2 performed in Sweden

Exclusion Criteria:

- Age below 18 years and 0 months at the time of transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Swedish citizens treated with ASCT for malignant disease in Sweden from 1st January 2020 until 31st December 2020 are eligible for this study. There will be a minimum follow-up time of one month for all patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 30 days
  Overall survival after infection with COVID-19
Overall survival | 90 days
  Overall survival after infection with COVID-19
COVID-19 related mortality | within 6 months after infection
  As classified by the WHO; a death resulting from a clinically compatible illness in a confirmed COVID-19 case, unless there is a clear alternative cause of death that cannot be related to COVID disease (e.g., trauma). There should be no period of complete recovery between the illness and death

SECONDARY OUTCOMES:
Time of COVID-19 infection | Up to 15 months
  Time of SARS-CoV-2 infection in relation to autologous stem cell transplantation
Hospitalization | Up to 15 months
  Duration of hospitalization
Oxygen treatment | Up to 15 months
  Duration of oxygen treatment
High-flow oxygen therapy | Up to 15 months
  Duration of high-flow oxygen therapy
Non-invasive ventilation | Up to 15 months
  Duration of non-invasive ventilation (NIV)
Intensive care | Up to 15 months
  Duration of care in intensive care unit
Invasive mechanical ventilation | Up to 15 months
  Duration of Invasive mechanical ventilation
ECMO | Up to 15 months
  Duration of extracorporeal membrane oxygenation (ECMO)
Occurence of ARDS | Up to 15 months
  Diagnosis of Acute respiratory distress syndrome (ARDS)
Occurence of arterial thrombosis | Up to 15 months
  Event of arterial thrombosis
Occurence of venous thrombosis | Up to 15 months
  Event of venous thrombosis
Occurence of arrhythmias | Up to 15 months
  Event of recorded arrhythmias
Occurence of acute cardiac injury | Up to 15 months
  Event of acute cardiac injury
Occurence of secondary infection | Up to 15 months
  Event of any secondary infection
Occurence of cytokine release syndrome | Up to 15 months
  Event of cytokine release syndrome
Comorbidities | Prior to autologous stem cell transplantation
  Description of comorbidities prior to autologous stem cell transplantation
Disease status | Prior to autologous stem cell transplantation
  Description of disease status prior to autologous stem cell transplantation
Previous disease modifying treatment | Prior to autologous stem cell transplantation
  Description of previous disease modifying treatment prior to autologous stem cell transplantation
Conditioning treatment | At autologous stem cell transplantation
  Description of conditioning treatment prior to autologous stem cell transplantation
Time of infection | At autologous stem cell transplantation or up to 15 months
  Time of COVID-19 in relation to autologous stem cell transplantation
Neutropenia | At autologous stem cell transplantation or up to 15 months
  Event of neutropenia at diagnosis of COVID-19
Elevated CRP | At autologous stem cell transplantation or up to 15 months
  Event of elevated C-reactive protein (CRP) at diagnosis of COVID-19
Elevated leukocyte count | At autologous stem cell transplantation or up to 15 months
  Event of elevated leukocyte count at diagnosis of COVID-19
Lymphocytopenia | At autologous stem cell transplantation or up to 15 months
  Event of lymphocytopenia at diagnosis of COVID-19
Elevated liver enzymes | At autologous stem cell transplantation or up to 15 months
  Event of elevated liver enzymes at diagnosis of COVID-19
Elevated lactate dehydrogenase | At autologous stem cell transplantation or up to 15 months
  Event of elevated lactate dehydrogenase at diagnosis of COVID-19
Elevated ferritin | At autologous stem cell transplantation or up to 15 months
  Event of elevated ferritin at diagnosis of COVID-19
Elevated d-dimer | At autologous stem cell transplantation or up to 15 months
  Event of elevated d-dimer at diagnosis of COVID-19
Prolonged aPTT | At autologous stem cell transplantation or up to 15 months
  Event of prolonged activated partial thromboplastin time (aPTT) at diagnosis of COVID-19
Elevated troponin | At autologous stem cell transplantation or up to 15 months
  Event of elevated troponin at diagnosis of COVID-19
Elevated creatinine | At autologous stem cell transplantation or up to 15 months
  Event of elevated creatinine at diagnosis of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Honar Cherif, MD, Ass prof, Principal Investigator — Department of Medical Sciences, Uppsala University; Thomas Silfverberg, MD, Study Chair — Center for Clinical Research Dalarna and Department of Medical Sciences-Uppsala University; Kristina Carlson, MD, Ass Prof, Study Chair — Department of Medical Sciences, Uppsala University
Locations (1):
- Uppsala Universitet, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Upon request the pseudonymized data sheet will be made available for other researchers depending on purpose of the request.

REFERENCES:
- [Background] Phelan AL, Katz R, Gostin LO. The Novel Coronavirus Originating in Wuhan, China: Challenges for Global Health Governance. JAMA. 2020 Feb 25;323(8):709-710. doi: 10.1001/jama.2020.1097. No abstract available. PMID 31999307
- [Background] Mossad SB, Longworth DL, Goormastic M, Serkey JM, Keys TF, Bolwell BJ. Early infectious complications in autologous bone marrow transplantation: a review of 219 patients. Bone Marrow Transplant. 1996 Aug;18(2):265-71. PMID 8864433
- [Background] Ljungman P, Ward KN, Crooks BN, Parker A, Martino R, Shaw PJ, Brinch L, Brune M, De La Camara R, Dekker A, Pauksen K, Russell N, Schwarer AP, Cordonnier C. Respiratory virus infections after stem cell transplantation: a prospective study from the Infectious Diseases Working Party of the European Group for Blood and Marrow Transplantation. Bone Marrow Transplant. 2001 Sep;28(5):479-84. doi: 10.1038/sj.bmt.1703139. PMID 11593321
- [Background] Hutspardol S, Essa M, Richardson S, Schechter T, Ali M, Krueger J, Fujii H, Egeler RM, Gassas A. Significant Transplantation-Related Mortality from Respiratory Virus Infections within the First One Hundred Days in Children after Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2015 Oct;21(10):1802-7. doi: 10.1016/j.bbmt.2015.06.015. Epub 2015 Jun 25. PMID 26117558
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Eichenberger EM, Soave R, Zappetti D, Small CB, Shore T, van Besien K, Douglass C, Westblade LF, Satlin MJ. Incidence, significance, and persistence of human coronavirus infection in hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2019 Jul;54(7):1058-1066. doi: 10.1038/s41409-018-0386-z. Epub 2018 Nov 1. PMID 30385869
- [Background] He W, Chen L, Chen L, Yuan G, Fang Y, Chen W, Wu D, Liang B, Lu X, Ma Y, Li L, Wang H, Chen Z, Li Q, Gale RP. COVID-19 in persons with haematological cancers. Leukemia. 2020 Jun;34(6):1637-1645. doi: 10.1038/s41375-020-0836-7. Epub 2020 Apr 24. PMID 32332856
- [Background] Ljungman P, Mikulska M, de la Camara R, Basak GW, Chabannon C, Corbacioglu S, Duarte R, Dolstra H, Lankester AC, Mohty M, Montoto S, Murray J, Peffault de Latour R, Snowden JA, Yakoub-Agha I, Verhoeven B, Kroger N, Styczynski J; European Society for Blood and Marrow Transplantation. The challenge of COVID-19 and hematopoietic cell transplantation; EBMT recommendations for management of hematopoietic cell transplant recipients, their donors, and patients undergoing CAR T-cell therapy. Bone Marrow Transplant. 2020 Nov;55(11):2071-2076. doi: 10.1038/s41409-020-0919-0. Epub 2020 May 13. PMID 32404975
- [Background] Terpos E, Engelhardt M, Cook G, Gay F, Mateos MV, Ntanasis-Stathopoulos I, van de Donk NWCJ, Avet-Loiseau H, Hajek R, Vangsted AJ, Ludwig H, Zweegman S, Moreau P, Einsele H, Boccadoro M, San Miguel J, Dimopoulos MA, Sonneveld P. Management of patients with multiple myeloma in the era of COVID-19 pandemic: a consensus paper from the European Myeloma Network (EMN). Leukemia. 2020 Aug;34(8):2000-2011. doi: 10.1038/s41375-020-0876-z. Epub 2020 May 22. PMID 32444866
- [Background] Dai M, Liu D, Liu M, Zhou F, Li G, Chen Z, Zhang Z, You H, Wu M, Zheng Q, Xiong Y, Xiong H, Wang C, Chen C, Xiong F, Zhang Y, Peng Y, Ge S, Zhen B, Yu T, Wang L, Wang H, Liu Y, Chen Y, Mei J, Gao X, Li Z, Gan L, He C, Li Z, Shi Y, Qi Y, Yang J, Tenen DG, Chai L, Mucci LA, Santillana M, Cai H. Patients with Cancer Appear More Vulnerable to SARS-CoV-2: A Multicenter Study during the COVID-19 Outbreak. Cancer Discov. 2020 Jun;10(6):783-791. doi: 10.1158/2159-8290.CD-20-0422. Epub 2020 Apr 28. PMID 32345594
- [Background] Pinana JL, Martino R, Garcia-Garcia I, Parody R, Morales MD, Benzo G, Gomez-Catalan I, Coll R, De La Fuente I, Luna A, Merchan B, Chinea A, de Miguel D, Serrano A, Perez C, Diaz C, Lopez JL, Saez AJ, Bailen R, Zudaire T, Martinez D, Jurado M, Calbacho M, Vazquez L, Garcia-Cadenas I, Fox L, Pimentel AI, Bautista G, Nieto A, Fernandez P, Vallejo JC, Solano C, Valero M, Espigado I, Saldana R, Sisinni L, Ribera JM, Jimenez MJ, Trabazo M, Gonzalez-Vicent M, Fernandez N, Talarn C, Montoya MC, Cedillo A, Sureda A; Infectious Complications Subcommittee of the Spanish Hematopoietic Stem Cell Transplantation and Cell Therapy Group (GETH). Risk factors and outcome of COVID-19 in patients with hematological malignancies. Exp Hematol Oncol. 2020 Aug 25;9:21. doi: 10.1186/s40164-020-00177-z. eCollection 2020. PMID 32864192
- [Background] Passamonti F, Cattaneo C, Arcaini L, Bruna R, Cavo M, Merli F, Angelucci E, Krampera M, Cairoli R, Della Porta MG, Fracchiolla N, Ladetto M, Gambacorti Passerini C, Salvini M, Marchetti M, Lemoli R, Molteni A, Busca A, Cuneo A, Romano A, Giuliani N, Galimberti S, Corso A, Morotti A, Falini B, Billio A, Gherlinzoni F, Visani G, Tisi MC, Tafuri A, Tosi P, Lanza F, Massaia M, Turrini M, Ferrara F, Gurrieri C, Vallisa D, Martelli M, Derenzini E, Guarini A, Conconi A, Cuccaro A, Cudillo L, Russo D, Ciambelli F, Scattolin AM, Luppi M, Selleri C, Ortu La Barbera E, Ferrandina C, Di Renzo N, Olivieri A, Bocchia M, Gentile M, Marchesi F, Musto P, Federici AB, Candoni A, Venditti A, Fava C, Pinto A, Galieni P, Rigacci L, Armiento D, Pane F, Oberti M, Zappasodi P, Visco C, Franchi M, Grossi PA, Bertu L, Corrao G, Pagano L, Corradini P; ITA-HEMA-COV Investigators. Clinical characteristics and risk factors associated with COVID-19 severity in patients with haematological malignancies in Italy: a retrospective, multicentre, cohort study. Lancet Haematol. 2020 Oct;7(10):e737-e745. doi: 10.1016/S2352-3026(20)30251-9. Epub 2020 Aug 13. PMID 32798473